CLINICAL TRIAL: NCT07083479
Title: Expanded Access Protocol for ELI-002 7P Immunotherapy as Treatment for Subjects With Kirsten Rat Sarcoma (KRAS)/Neuroblastoma RAS Viral Oncogene Homolog (NRAS) Mutated Pancreatic Ductal Adenocarcinoma (PDAC)
Brief Title: Expanded Access Protocol of ELI-002-102 in Subjects With KRAS/NRAS Mutated Pancreatic Ductal Adenocarcinoma
Acronym: AMPLIFY-EAP
Status: Available | Type: Expanded Access
Sponsor: Elicio Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: ELI-002-102
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Ductal Adenocarcinoma; KRAS G12D; KRAS G12V; KRAS G12S; KRAS G12A; KRAS G12C; KRAS G12R; KRAS G13D; NRAS G12D; NRAS G12V; NRAS G12S; NRAS G12A; NRAS G12C; NRAS G12R; NRAS G13D
Keywords: Pancreatic ductal adenocarcinoma (PDAC); Kirsten rat sarcoma (KRAS); Neuroblastoma ras viral oncogene homolog (NRAS); Adjuvant therapy; Immunotherapy; Vaccine therapy; Expanded access; Expandd access protocol (EAP)

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: ELI-002 7P — ELI-002 Amph-CpG-7909 (10.0 mg) admixed with ELI-002 Amph-Peptides 7P (4.9 mg) administered via SC injection weekly for 4 consecutive weeks, followed by bi-weekly injections over 4 weeks, during the Immunization Period; additional SC injections weekly for 4 weeks during the Booster Period (the two periods are separated by 2 months of no dosing).

SUMMARY:
This is an open-label expanded access protocol (EAP) of ELI-002 7P immunotherapy (a lipid-conjugated immune-stimulatory oligonucleotide [Amph-CpG-7909] plus a mixture of lipid-conjugated peptide-based antigens [Amph-Peptides 7P]) as adjuvant treatment in patients with KRAS/NRAS-mutated pancreatic ductal adenocarcinoma who are at high risk for relapse (ie, presence of isolated tumor cells in a patient whose primary tumor has been removed and is currently without clinical signs of disease). This protocol builds on the experience being obtained with ELI-002 7P (with Amph-Peptides G12D, G12R, G12V, G12A, G12C, G12S, G13D), which is being studied in protocol ELI-002-201.

DETAILED DESCRIPTION:
This EAP was designed to provide ELI-002 7P access to patients when all of the following apply: patient has a serious or immediately life-threatening disease or condition; there is no comparable or satisfactory alternative therapy to diagnose, monitor, or treat the disease or condition; patient enrollment in a clinical trial is not possible; potential patient benefit justifies the potential risks of treatment; and providing the investigational medical product will not interfere with investigational trials that could support a medical product's development or marketing approval for the treatment indication. In addition, the protocol will include patients participating in Study ELI-002-201 who might benefit from receiving doses beyond the protocol-specified schedule for that study. As such, this EAP will include 2 cohorts: Cohort 1A will include patients unable to participate in other clinical trial protocols and will receive ELI-002 7P for the first time; and Cohort 1B will include patients who have completed the dosing specified in Study ELI-002-201 and are receiving additional booster doses.

The protocol consists of a Screening Period, an Immunization Period, a 2-Month No Dosing Period, a Booster Period, and a Follow-up Period. Patients who have not previously received ELI-002 7P (Cohort 1A) will participate in all periods of the protocol. Patients who have completed previous treatment with ELI-002 7P and are only receiving additional booster doses (Cohort 1B) will skip the Immunization Period and 2-Month No Dosing Period. All patients will receive booster doses unless they have unresolved toxicity (specific to Cohort 1A).

All patients will be observed for safety and tolerability. Laboratory assessments (hematology, blood chemistry), vital signs, physical examinations, and radiographic imaging and other assessments will be performed per institution standard of care practice and per treating physician judgement. Patients with confirmed radiographic relapse (using iRECIST criteria; not judged as pseudoprogression) during treatment with ELI-002 7P may either discontinue trial treatment or continue trial treatment if the treating physician determines that continued use of ELI-002 7P is appropriate treatment for the current clinical situation, the patient is tolerating ELI-002 7P, and the patient has stable performance status.

ELIGIBILITY:
Inclusion Criteria:

* Has at least 1 of the 7 KRAS/NRAS mutated alleles (G12D, G12R, G12V, G12A, G12C, G12S, G13D)
* The following must be met: (1) the patient has no alternative therapy to diagnose, monitor, or treat the disease or condition; (2) enrollment in a clinical trial is not possible; and (3) the potential benefit to the patient justifies the potential risks of treatment.
* Screening CT scan negative for recurrent disease
* Eastern Cooperative Oncology Group performance status of 0 or 1

Exclusion Criteria:

* Use of immunosuppressive drugs
* Known brain metastases

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult